CLINICAL TRIAL: NCT02679586
Title: Evaluation of an Imaging Biomarker for Early Detection of Treatment Efficacy During Breast Cancer Neoadjuvant Chemotherapy
Brief Title: Imaging Biomarker for Early Detection of Treatment Efficacy During Breast Cancer Neoadjuvant Chemotherapy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Principal Investigator, Lynn Henry, Associate Professor of Internal Medicine, University of Michigan Rogel Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UMCC 2006.010; HUM00003392 (Other: University of Michigan)
Record Dates: First submitted 2016-02-05; First posted 2016-02-10 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Diffusion Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diffusion weighted MRI Group (Experimental): All patients will receive a double baseline diffusion weighted MRI (performed on the same day as the Baseline MRI).
  Patients participating in Part I will receive another MRI approximately 1 week (day 8-11) after the first dose of Chemotherapy (chemotherapy will be determined by the treating physician and is not assigned as part of this trial).
  Patients participating in Part II will receive a single MRI 1-2 weeks after the first dose of Chemotherapy A (chemotherapy will be determined by the treating physician and is not assigned as part of this trial). A second MRI will be repeated within 2 weeks prior to the start of Chemotherapy B.
  Interventions: Device: Diffusion weighted MRI

INTERVENTIONS:
Device: Diffusion weighted MRI
  Other Names: DW-MRI

SUMMARY:
This is a single-arm, single-institution pilot study that will collect preliminary data to be used in the design of a subsequent study to assess whether changes in fDM (Functional Diffusion Maps) derived from primary breast cancer diffusion weighted MRI images can serve as an early predictor of response to treatment, and whether the magnitude of the change correlates with the effectiveness of treatment.

DETAILED DESCRIPTION:
This trial has a two-step, sequential design, with continuation to the second part of the trial being dependent on the positive results in the first part. In Part One of the trial, the investigator will compare intrapatient variability in fDM performed at two timepoints prior to chemotherapy (chemotherapy will be chosen by the treating physician and will not be assigned as part of this study), with the change in fDM before and approximately one week after a dose of chemotherapy, to establish that treatment-related changes in fDM will occur in this clinical setting. If there are positive results in Part One, then the investigator will proceed to the second half of the trial. In Part Two, the investigator will examine changes in fDM that occur one week after each type of chemotherapy is administered, which will be compared to pathologic response, radiological response, and clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a primary measurable, biopsy proven, invasive breast carcinoma with the primary tumor intact. The tumor should be staged clinically as T2-T4 (minimum size >2.0 cm).
* Patients must have a breast tumor that is resectable or potentially resectable following neoadjuvant chemotherapy and be willing to undergo resection, if indicated, after chemotherapy.
* Patients may not have received prior chemotherapy or radiation therapy for their current breast cancer.
* Patients may not have had a clip placed into the tumor that is not compatible with MRI.
* Patients must be deemed eligible for neoadjuvant chemotherapy, as assessed by the clinical investigator.
* Age > 18 years.
* Patients must have an ECOG performance status (Eastern Cooperative Oncology Group Performance Status: an attempt to quantify cancer patients' general well-being and activities of daily life. The score ranges from 0 to 5 where 0 is asymptomatic and 5 is death.) of 0 - 1.
* Patients must not be pregnant or breast-feeding. Patients with reproductive potential must consent to the use of effective contraception while on the study.
* Patients must have no contraindications to MRI (Magnetic Resonance Imaging) exams. Patients who require sedation with general anesthesia to complete an MRI are not eligible for the study.
* Patients may have no ferrous metal implants or medical devices which would exclude MRI.
* Patients must be capable of lying flat in an MRI magnet for 30-60 minutes on 4 occasions.
* Weight must be less than 275 pounds.
* Patients must have the ability to understand and willingness to sign a written informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-06; Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Percent change in apparent diffusion coefficient between baseline and 8-11 days after chemotherapy | baseline and 8-11 days post treatment
  Percent change in apparent diffusion coefficient was determined by calculating the percentage change between the value prior to chemotherapy and at 8-11 days post treatment for treatment responders (patients with Complete Response [CR] or Partial Response [PR]) and for the treatment non-responders (patients with Stable Disease [SD] or Progressive Disease [PD]).

SECONDARY OUTCOMES:
Change in relative tumor volume with increasing apparent diffusion coefficient between baseline and 8-11 days of chemotherapy | baseline and 8-11 days post treatment
  Determine, by Parametric Response Map (PRM), the percent relative tumor volume with increasing ADC in responders (patients with Complete Response [CR] or Partial Response [PR]) and non-responders (patients with Stable Disease [SD] or Progressive Disease [PD].
Change in relative tumor volume with decreasing apparent diffusion coefficient between baseline and 8-11 days of chemotherapy | baseline and 8-11 days post treatment
  Determine, by Parametric Response Map (PRM), the percent relative tumor volume with decreasing ADC in responders (patients with Complete Response [CR] or Partial Response [PR]) and non-responders (patients with Stable Disease [SD] or Progressive Disease [PD].

CONTACTS AND LOCATIONS:
Overall Officials: Norah L Henry, M.D., Ph.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Galban CJ, Ma B, Malyarenko D, Pickles MD, Heist K, Henry NL, Schott AF, Neal CH, Hylton NM, Rehemtulla A, Johnson TD, Meyer CR, Chenevert TL, Turnbull LW, Ross BD. Multi-site clinical evaluation of DW-MRI as a treatment response metric for breast cancer patients undergoing neoadjuvant chemotherapy. PLoS One. 2015 Mar 27;10(3):e0122151. doi: 10.1371/journal.pone.0122151. eCollection 2015. PMID 25816249